CLINICAL TRIAL: NCT01574924
Title: Personality Change During Medical Residency Across Different Medical Specialties
Brief Title: Personality Change During Medical Residency
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Coimbra (Other)
Responsible Party: Principal Investigator, Fernanda Cristina Ordens Miguel, MD, University of Coimbra
Other Study IDs: PERINT-01
Record Dates: First submitted 2012-04-05; First posted 2012-04-10 (Estimated); Last update posted 2012-04-16 (Estimated); Status verified 2012-04

CONDITIONS: Personality; Coping Skills
Keywords: Personality change; Perfectionism; Coping; Medical Specialty; Medical Residency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Medical residents
  Interventions: Other: No intervention.

INTERVENTIONS:
Other: No intervention. — There are no interventions in this observational study.

SUMMARY:
The Ethics Committee of Hospital and University Center of Coimbra (Portugal) complies, reports and is supervisioned by the Portuguese Ethics Committee.

The Ethics Committee of Hospital and University Center of Coimbra is an multidisciplinary organ of Ethics experts that give support to the board of hospital directors, the health personnel and patients, regarding bioethical issues emerging from clinical assistance activities (addressed to patient's health being, education and clinical research).

ELIGIBILITY:
Inclusion Criteria:

* Medical residents with ages between 23 and 45 years old, attending the first year of medical specialty in Portugal in the following specialties*: General Surgery, Neurosurgery; Orthopedics; Intern Medicine, Gastroenterology; Cardiology; Rheumatology; Endocrinology; Oncology; Intensive Medicine; Pediatric; Radiology; Clinical Pathology; Neurology and Psychiatry.
* Acceptance and commitment to participate in the study.
* Signature of study' informed consent.

Exclusion Criteria:

* Attendance, during the study, in an international formative stage with a duration superior to 12 months.
* Previous attendance of other medical specialty for more than one year.
* Present or past history of major psychiatry disorders (illicit drug abuse with dependence, schizophrenia, bipolar disorder or schizoaffective disorder)

Ages: 23 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: All portuguese medical (first year) residents will be invited to participate in the study (target population).
  Targeted enrollment stategies will be used to recruit participants (individual invitation emails). Also, the study will be disclosed in some social networks. The research team has created a proper email account (personalidade.internato@gmail.com) to answer any questions and to change email with the participants of the study.
  To those who accepted and consent to participate (study population), it will be send the online link to create a confidential account and access (and to give answers to the questionnaires).
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2012-04; Primary Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Personality | First assessment: 1st month of medical specialty. Second (final) assessment: 1st month after medical specialty final exam [4, 5, 6 (or more) years after the 1st evaluation, according to the time taken to complete medical residency].
  Change in the facets of personality domains (Neuroticism, Extroversion and Conscientiousness) measure with the portuguese version (Lima et al) of NEO PI-R (Costa & McCrae).

SECONDARY OUTCOMES:
Perfectionism | First assessment: 1st month of medical specialty. Second (final) assessment: 1st month after medical specialty final exam [4, 5, 6 (or more) years after the 1st evaluation, according to the time taken to complete medical residency].
  Baseline (and changes)in Perfectionism measured using the portuguese version (Soares et al) of Multidimensional Perfectionism Scale (Frost)
Problem Solving Inventory (Vaz Serra et al) | First assessment: 1st month of medical specialty. Second (final) assessment: 1st month after medical specialty final exam [4, 5, 6 (or more) years after the 1st evaluation, according to the time taken to complete medical residency].

CONTACTS AND LOCATIONS:
Overall Officials: Fernanda Miguel, MD, Principal Investigator — Department of Psychiatry at Hospital and University Center of Coimbra, EPE; Fernanda Miguel, MD, Study Chair — Department of Psychiatry at Hospital and University Center of Coimbra, EPE; Eva Mendes, MD, Study Chair — Department of Psychiatry at Hospital and University Center of Coimbra, EPE; Susana Renca, MD, Study Chair — Department of Psychiatry at Hospital and University Center of Coimbra, EPE; Joana Andrade, MD, Study Chair — Department of Psychiatry at Hospital and University Center of Coimbra, EPE; Sandra Pereira, MD, Study Chair — Department of Psychiatry at Hospital and University Center of Coimbra, EPE; Catarina Pereira, MD, Study Chair — Department of Psychiatry at Hospital and University Center of Coimbra, EPE; Helena Rita, MD, Study Chair — Department of Psychiatry at Hospital and University Center of Coimbra, EPE; Joaquim Cerejeira, MD. Ph D, Study Chair — Department of Psychiatry at Hospital and University Center of Coimbra, EPE; Ana Cabral, MD, Study Chair — Department of Psychiatry at Hospital and University Center of Coimbra, EPE; Salomé Caldeira, Clinical Psychologist, Study Chair — Department of Psychiatry at Hospital and University Center of Coimbra, EPE; Maria Soares, Ph D, Study Chair — Institute of Medical Psychology, Faculty of Medicine, University of Coimbra; Telma Pereira, PhD, Study Chair — Institute of Medical Psychology, Faculty of Medicine, University of Coimbra; António Macedo, MD. PhD, Study Director — Institute of Medical Psychology, Faculty of Medicine, University of Coimbra; Department of Psychiatry at Hospital and University Center of Coimbra, EPE
Locations (1):
- Department of Psychiatry at Hospitalar and Universitary Center of Coimbra, EPE, Coimbra, Portugal